CLINICAL TRIAL: NCT00286546
Title: The Role of Testosterone in Major Depression
Brief Title: Testosterone and Major Depression
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: 002
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2005-08

CONDITIONS: Major Depression
Keywords: Testosterone; Major Depression; Men
MeSH Terms: conditions — Depressive Disorder, Major; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Context - As men age, testosterone levels decline leading to symptoms that overlap with the symptoms of major depression. Little is known about the potential role of testosterone in the treatment of major depression.Objective - To assess the levels of bioavailable testosterone and total levels of testosterone in men diagnosed with major depressive disorder between the ages of 40 and 65.Design, Setting and Participants - 50 men between the ages of 40 and 65 and who suffer from major depressive disorder will be compared with 50 age matched healthy controls in an outpatient hospital setting. Main Outcome Measures - Bioavailable testosterone and total testosterone levels will be measured as well as blood pressure, pulse rate, height, weight, waist and hip measurements. Medical and psychiatric history will be assessed by the study physician. The Mini International Neuropsychiatric Interview (MINI) will be used to administered by the physician to ensure that the patient meets the DSM-IV criteria for Major Depression. The Hamilton Depression Rating Scale (HAM-D-17) will be used to assess depression symptom severity. A Symptom/Side Effect Rating Scale will also be administered to measure the presence and severity of side effects that each patient may be experiencing. In addition, the SEX FX questionnaire will be administered. Each patient will be asked to complete a series of self-report measures including the Social Adaptation Self-Evaluation Scale Questionnaire (SASS), the Androgen Deficiency in Aging Males (ADAM) and the Beck Depression Inventory (BDI-II).

DETAILED DESCRIPTION:
This study will be carried our at the Mood Disorders Psychopharmacology Unit (MDPU), University Health Network (UHN), University of Toronto, with the approval of the Research Ethics Board (REB). Informed consent will be obtained from all subjects prior to study enrollment.50 male subjects between the age of 40 and 65 will be evaluated by the psychiatrist to assess whether each patient meets DSM-IV criteria for Major Depression using the MINI and to obtain their medical and psychiatric history. In addition, the SEX FX questionnaire (an instrument measuring sexual dysfunction) will be administered. Once each patient has signed the informed consent document, the research staff will assess the severity of depressive symptoms by administering the Hamilton Depression Rating Scale (HAM-D-17). A Symptom/Side Effect Rating Scale will also be administered to measure the presence and severity of side effects that each patient may be experiencing. Each patient will then have pulse, blood pressure, weight, height, waist and hip measurements taken to evaluate their health. Patients will be asked to provide blood (about 3 teaspoons) and urine (about 1/4 cup) samples for laboratory tests (bioavailable testosterone, LH, thyroid and prolactin). The blood samples will be obtained in the morning between 0800 and 1100 hr. Each patient will then be asked to complete a series of self-report measures including the SASS, the ADAM, and the Beck Depression Inventory.The 50 healthy controls will have a structured diagnostic interview (MINI) administered by the coordinator to obtain their psychiatric and medical history. They will undergo all laboratory tests required of the depressed population and all rating scales mentioned above will be completed with this population as well. Each patient is free to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM IV criteria for a diagnosis of Major Depressive Disorder as per an assessment by the PREN physician-investigator.
* Subjects must have a Hamilton Depression Rating Scale (HAM-D-17) of at least 16.
* Subjects must be male between the ages of 40 and 65.
* Subjects must be judged by the investigator to be in generally good health.
* Body Mass Index (BMI) between 20 to 29 kg/m2.
* Able and willing to give meaningful written consent.
* Educational level and a degree of understanding such that they can communicate effectively with the Investigator.
* Subjects must have had normal sexual functioning prior to the onset of depression.

Exclusion Criteria:

* Subjects must not suffer from clinically significant medical conditions. Examples include neurological, cardiovascular, gastrointestinal, hepatic, renal, haematological, respiratory or endocrine illnesses.
* Recent history of drug or alcohol abuse/dependence within the past 6 months as defined by DSM-IV or in the opinion of the investigator.
* Uncorrected hypothyroidism or hyperthyroidism.
* Current use of hormone replacement therapy.
* Current diagnosis of schizophrenia or other psychotic disorder (including psychotic disorder due to general medical condition, substance-induced psychotic disorder, psychotic disorder not otherwise specified) as defined in the DSM-IV.
* Current diagnosis of depressive disorder not otherwise specified or bipolar I disorder, most recent episode major depression mixed or manic bipolar II disorder as defined in the DSM-IV.
* Electroconvulsive therapy (ECT) within the 3 months prior to visit 1.
* Not currently on any antidepressants or must have an interval of the following prior to entry into the study: Fluoxetine-4 weeks; MAOIs- 2 weeks
* All other psychotic medications and herbal preparations with putative antidepressant properties (e.g. paroxetine HCI, other antidepressant not specified above, St. John's Wort, kava-kava or Valerian: 1 week)

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-01; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Roger McIntyre, MD, FRCPC, Principal Investigator — University Health Network, University of Toronto; Roger McIntyre, Principal Investigator — UHN Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada